CLINICAL TRIAL: NCT03416270
Title: ERtugliflozin triAl in DIabetes With Preserved or Reduced ejeCtion FrAcTion mEchanistic Evaluation in Heart Failure: "ERADICATE-HF"
Brief Title: ERtugliflozin triAl in DIabetes With Preserved or Reduced ejeCtion FrAcTion mEchanistic Evaluation in Heart Failure
Acronym: ERADICATE-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University Medical Center Groningen (Other); Merck Sharp & Dohme LLC (Industry); University of Toronto (Other); Toronto General Hospital (Other)
Responsible Party: Principal Investigator, David Z.I. Cherney, Associate Professor of Medicine, Clinician Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-5627
Record Dates: First submitted 2018-01-15; First posted 2018-01-31 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes Mellitus; Heart Failure
Keywords: SGLT2 inhibtion; Ertugliflozin; Type 2 Diabetes; Heart Failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure | interventions — ertugliflozin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to 15 mg (10mg + 5mg tablets) PO ertugliflozin daily or a matched placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ertuglifozin Treatment Arm (Experimental): Ertugliflozin Tablets Total Dose 15mg (10mg + 5 mg) for 12 weeks
  Interventions: Drug: Ertugliflozin
- Placebo Arm (Placebo Comparator): Placebo Matching Ertugliflozin Tablet for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ertugliflozin — Ertugliflozin Tablets Total Dose 15mg (10mg + 5 mg) once daily for 12 weeks
  Arms: Ertuglifozin Treatment Arm
Drug: Placebo — Placebo once daily for 12 weeks
  Arms: Placebo Arm

SUMMARY:
This study aims to elucidate the mechanisms whereby the SGLT2i "ertugliflozin" modifies cardiorenal interactions that regulate fluid volume and neurohormonal activation in patients with type 2 diabetes and heart failure (T2D-HF).

DETAILED DESCRIPTION:
Newer agents called sodium glucose co-transporter-2 inhibitors (SGLT2i) have been developed to improve glycemic control and lower hemoglobin A1c by increasing glycosuria. SGLT2i also reduce blood pressure and albuminuria in T2D - possibly through natriuresis. Importantly, a landmark trial "EMPA-REG OUTCOME" demonstrated that the SGLT2i "empagliflozin" is the first anti- hyperglycemic agent to reduce mortality and HF risk, and also to decrease the risk of progressive diabetic nephropathy. Similar benefits were also recently reported in the CANVAS Program trial with canagliflozin. Despite the benefits observed in these two pivotal trials, the mechanisms responsible for beneficial effects of SGLT2i in patients with T2D with respect to the development and/or worsening of HF are not currently known.

In light of the results of EMPA-REG OUTCOME, the investigators aim to elucidate the mechanisms whereby the SGLT2i "ertugliflozin" modifies cardiorenal interactions that regulate fluid volume and neurohormonal activation in patients with T2D and HF (T2D-HF). The investigators will test the hypothesis that ertugliflozin increases proximal tubular natriuresis, thereby reducing plasma volume, without inducing significant renal vasoconstriction or activation of the sympathetic nervous system (SNS) (see below, Figure 1). The systematic understanding of the effects of SGLT2i in the setting of HF will enable the design of rational physiology based strategies to decrease the burden of HF, which could have major clinical and research implications internationally.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects diagnosed with T2D ≥12 months prior to informed consent;
2. eGFR ≥30 ml/min/1.73m2;
3. Age >18 years;
4. HbA1c 6.5%-10.5%;
5. Body Mass Index (BMI) 18.5-45.0 kg/m2;
6. Blood pressure ≤160/110 and ≥90/60 at screening,
7. Heart failure with New York Heart Association (NYHA) class 2-3 symptoms and ejection fraction ≥20%
8. Stable dose of maximally tolerated ACE inhibitor, angiotensin receptor blocker or renin inhibitor for at least 30 days
9. Stable diuretic dose for at least 30 days at the time of baseline physiological assessment
10. BNP levels at baseline ≥100 pg/ml (no atrial fibrillation), ≥200 pg/ml if in atrial fibrillation

Exclusion Criteria:

1. Type 1 Diabetes;
2. Leukocyte and/or nitrite positive urinalysis that is untreated;
3. Severe hypoglycaemia within 2 months prior to screening;
4. History of brittle diabetes or hypoglycaemia unawareness based on investigator judgement;
5. Unstable coronary artery disease with acute coronary syndrome, percutaneous intervention or bypass surgery within 3 months;
6. Clinically significant valvular disease;
7. Congestive heart failure secondary to an infiltrative cardiomyopathic process (for example amyloid) or pericardial constriction;
8. Uncontrolled systemic hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >110) or systemic hypotension (systolic blood pressure < 90/60 mmHg);
9. Bariatric surgery or other surgeries that induce chronic malabsorption;
10. Anti-obesity drugs or diet regimen and unstable body weight three months prior to screening;
11. Treatment with systemic corticosteroids;
12. Blood dyscrasias or any disorders causing hemolysis or unstable red blood cells;
13. Pre-menopausal women who are nursing, pregnant, or of child-bearing potential and not practicing an acceptable method of birth control;
14. Participation in another trial with an investigational drug within 30 days of informed consent;
15. Alcohol or drug abuse within three months prior to informed consent that would interfere with trial participation or any ongoing clinical condition that would jeopardize subject safety or study compliance based on investigator judgement;
16. Liver disease, defined by serum levels of alanine transaminase, aspartate transaminase, or alkaline phosphatase >3 x upper limit of normal as determined during screening;
17. Active malignancy at the time of screening;

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David ZI Cherney, MD PhD, Principal Investigator — University Health Network, Toronto General Hospital
Locations (3):
- Toronto General Hospital, Toronto, Ontario, Canada
- Netherlands (2):
  - Vanderbilt University Medical Centre, Amsterdam, De Boelelaan
  - University Medical Center Groningen, Groningen

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Started | 17 | 17
Completed | 17 | 16
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (8.7) | 69.4 (7.5) | 69.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 15 | 13 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 13 | 12 | 25
  Black | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Other | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 8 | 16
  Netherlands | 9 | 9 | 18
eGFR [Mean (Standard Deviation); unit: mL/min/1.73 m2] | 63.5 (23.3) | 66.4 (22.4) | 65 (22.9)

OUTCOME MEASURES:

1. Primary Outcome: Fractional Excretion of Lithium (FELi)
Description: The difference in fractional excretion of lithium (FELi) with ertugliflozin vs. placebo. This was measured using exogenous lithium administration 12 hours before lithium excretion was measured in urine and blood.
Time Frame: Change in outcomes was measured acute (1 week minus baseline values) and chronic (12 weeks minus baseline values)
Measure: Mean (Standard Error); unit: percentage of filtered lithium excreted
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
percentage of filtered lithium excreted
  Week 1 | 0.3 (6.9) | -2.3 (16.8)
  Week 12 | 0.8 (11.0) | -4.9 (16.6)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.36, Wilcoxon (Mann-Whitney) — 12 weeks
Statistical Analysis 2: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.56, Wilcoxon (Mann-Whitney) — 1 week

2. Secondary Outcome: Glomerular Filtration Rate (GFR)
Description: The difference in iohexol-measured GFR with ertugliflozin vs. placebo. 5ml bolus iohexol (Omnipaque 300mg) was infused intravenously over 2 minutes while participants were supine. Iohexol disappearance curve was used to measure GFR over from 2-4 hours after infusion.
Time Frame: Glomerular Filtration Rate (GFR, based on plasma iohexol clearance) will be measured at 12 weeks
Measure: Mean (Standard Error); unit: mL/min/1.73 m2
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
mL/min/1.73 m2 | 48.6 (4.0) | 50.1 (4.2)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.303, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Effective Renal Plasma Flow (ERPF)
Description: The difference in ERPF with ertugliflozin vs. placebo. Paraaminohippurate (PAH) was intravenously administered to measured ERPF.
Time Frame: Effective Renal Plasma Flow (ERPF, based on paraaminohippurate plasma clearance) will be measured at 12 weeks
Measure: Mean (Standard Error); unit: mL/min/1.73 m2
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
mL/min/1.73 m2 | 399.1 (46.8) | 335.6 (41.5)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.438, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: The difference in seated SBP with ertugliflozin vs. placebo
Time Frame: chronic (12 weeks)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
mmHg | 132 (5) | 128 (5)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.599, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: The difference in seated DBP with ertugliflozin vs. placebo
Time Frame: chronic (12 weeks)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
mmHg | 77 (3) | 76 (3)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.92, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Heart Rate (HR)
Description: The difference in seated HR with ertugliflozin vs. placebo
Time Frame: chronic (12 weeks)
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
bpm | 74 (3) | 72 (3)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.405, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: LV Ejection Fraction
Description: Echocardiography for markers of systolic and diastolic function
Time Frame: chronic (12 weeks)
Measure: Mean (Standard Error); unit: percentage of output
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
percentage of output | 49.2 (4.4) | 43.6 (5.4)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.536, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Carotid-femoral Pulse Wave Velocity
Description: Arterial Stiffness using SphygmaCor software. Pulse points measured at carotid and femoral arteries.
Time Frame: chronic (12 weeks)
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
m/s | 11.50 (1.50) | 12.14 (1.42)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.443, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Plasma Volume
Description: Plasma volume will be measured using a non-radioactive technique (indocyanine green dilution)
Time Frame: chronic (12 weeks)
Population: The plasma volume was calculated from the laboratory-measured indocyanine green dye values in n=18 participants who had measurements performed.
Measure: Mean (Standard Error); unit: ml
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 9 | 9
ml | 3470.9 (438) | 3158.2 (491.9)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.849, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Extracellular Water
Description: Extracellular water will be measured non-invasively using bioimpedence spectroscopy
Time Frame: chronic (12 weeks)
Measure: Mean (Standard Error); unit: L
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
L | 20.1 (0.9) | 21.8 (1.0)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.013, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Cardiac Output
Description: Cardiac output will also be measured using non-invasive cardiac monitoring (NICOM)
Time Frame: chronic (12 weeks)
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
L/min | 5.8 (0.3) | 5.8 (0.3)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.844, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Systemic Vascular Resistance
Description: Systemic vascular resistance will also be measured using non-invasive cardiac monitoring (NICOM)
Time Frame: chronic (12 weeks)
Measure: Mean (Standard Error); unit: dynes·s·cm5
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
dynes·s·cm5 | 1346.7 (99.1) | 1437.1 (99.9)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.262, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Blood Angiotensin II
Description: Neurohormones/biomarkers
Time Frame: chronic (12 weeks)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
pg/ml | 89.2 (7.1) | 86.5 (7.3)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.802, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: BNP
Description: Neurohormones/biomarkers
Time Frame: chronic (12 weeks)
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
pg/ml | 1311.1 (400.5) | 576.6 (405.3)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.327, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Norepinephrine
Description: Neurohormones/biomarkers
Time Frame: chronic (12 weeks)
Measure: Mean (Standard Error); unit: nM
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
nM | 2.6 (0.3) | 2.6 (0.3)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.618, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Urinary Adenosine
Description: Neurohormones/biomarkers
Time Frame: chronic (12 weeks)
Measure: Mean (Standard Error); unit: mM/μmol Cr
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
mM/μmol Cr | 0.25 (0.05) | 0.39 (0.05)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm; Test type: Other; p = 0.946, Wilcoxon (Mann-Whitney)

17. Primary Outcome: Fractional Excretion of Sodium (FENa)
Description: The difference in fractional excretion of sodium (FENa) with ertugliflozin vs. placebo. This was measured using exogenous lithium administration 12 hours before sodium excretion was measured in urine and blood.
Time Frame: Change in outcomes was measured acute (1 week minus baseline values) and chronic (12 weeks minus baseline values)
Measure: Mean (Standard Error); unit: percentage of sodium excretion
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
percentage of sodium excretion
  Week 1 | -0.6 (1.9) | 0.3 (1.7)
  Week 12 | -0.6 (1.6) | 0.1 (1.3)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.53, Wilcoxon (Mann-Whitney) — 12 week
Statistical Analysis 2: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.89, Wilcoxon (Mann-Whitney) — 1 week

18. Primary Outcome: Change in Absolute Fractional Distal Sodium Reabsorption From Baseline (FELi-FENa)
Description: The difference in fractional excretion of lithium and fractional excretion of sodium (calculated by the difference between FELi and FENa) with ertugliflozin vs. placebo. This was measured using exogenous lithium administration 12 hours before sodium excretion was measured in urine and blood.
Time Frame: Change in outcomes was measured acute (1 week minus baseline values) and chronic (12 weeks minus baseline values)
Measure: Mean (Standard Error); unit: percentage of total sodium reabsorption
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
Number analyzed (Participants) | 17 | 16
percentage of total sodium reabsorption
  Week 1 | 0.8 (7.0) | -2.6 (16.7)
  Week 12 | 1.4 (10.6) | -5 (16.1)
Statistical Analysis 1: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.26, Wilcoxon (Mann-Whitney) — 12 weeks
Statistical Analysis 2: Comparison: Ertuglifozin Treatment Arm vs Placebo Arm; Test type: Other; p = 0.56, Wilcoxon (Mann-Whitney) — 1 week

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Ertuglifozin Treatment Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 3/17 | 1/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertuglifozin Treatment Arm (N=17) | Placebo Arm (N=17)
Heart failure hospitalization (Cardiac disorders) | 1 (3) | 0 (0)
Emesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
There are limitations to the present analysis. Due to increasing use of SGLT2 inhibition for the clinical indication of HF and challenges posed by the COVID-19 pandemic, we were unable to meet the participant recruitment target for this trial. Therefore, our study was potentially underpowered to detect a difference between ertugliflozin and placebo groups in the primary outcome of FELi.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT03416270/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT03416270/SAP_001.pdf